CLINICAL TRIAL: NCT00839462
Title: Evaluation of the Effect of Bepanthen Burn Relief Foam Spray New Formula on a Thermic Erythema. Equivalence Trial. Intra-individual Design.
Brief Title: Efficacy of Dexpanthenol in Thermic Erythema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12039
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Erythema
Keywords: Thermal Erythema; Dexpanthenol; Erythema; Efficacy
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Dexpanthenol foam spray, new formulation
- Arm 2 (Active Comparator)
  Interventions: Drug: Dexpanthenol foam spray, old formulation

INTERVENTIONS:
Drug: Dexpanthenol foam spray, new formulation — 2 applications of 2 micro liter/square centimeter on a 4X4 cm area corresponding to 32 micro liter
  Arms: Arm 1
Drug: Dexpanthenol foam spray, old formulation — 2 applications of 2 micro liter/square centimeter on a 4X4 cm area corresponding to 32 micro liter
  Arms: Arm 2

SUMMARY:
The study focuses to prove the equivalent efficacy of two different Dexpanthenol formulations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Phototype: I to IV according to Fitzpatrick scale

Exclusion Criteria:

* Pregnant or nursing women
* Subjects registered as being in exclusion period in the French Health Minister file of subjects
* Subjects with known allergy to cosmetics, skin care products, or topical drugs, a sensitivity related to any component of any formulations being tested

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Global sum of scores for evaluating the cooling/soothing effect evaluated after first and second application | 2 min, 5 min, 10 min, 15 min

SECONDARY OUTCOMES:
Skin temperature | 2 min, 5 min, 10 min
Evaluation of the cooling/soothing effect (scores) after first and second application | 2 min, 5min, 10 min, 15 min
Evaluation of the foam covering properties after first application | 2 min, 5 min, 10 min, 15 min
Incidence of adverse events | FPFV - LPLV

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Villeurbanne, France